CLINICAL TRIAL: NCT06324552
Title: Defects of Keratinocytes Function in Dermatologic Patients Carrying Genetic Variants Involved in NOTCH Signaling
Brief Title: Defects of Keratinocytes Function in Dermatologic Patients
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 16/18
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; NOTCH signaling
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
NOTCH signaling in the skin exerts a pivotal role in the regulation of normal keratinocytes turnover by mediating the balance between proliferation, differentiation, apoptosis and autophagic flux progression. Two skin diseases are characterized by the presence of gene variants that cause an impairment in NOTCH signaling: hidradenitis suppurativa(HS) and Dowling-Degos disease(DDD). To date, both HS and DDD are orphan diseases still lacking of specific treatments. This project aims at improving the current knowledge on the pathogenesis of HS and DDD, by deepening the understandings on the role played by keratinocytes in these pathologies and also by determining why mutations found in the same pathway cause different diseases. This study aimed to obtain in vitro models, derived directly from patients (from hair follicles) and from keratinocytes (HaCaT) cell cultures, for the study of these skin pathologies and also for the testing of novel innovative therapies such as photobiomodulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of HS

Exclusion Criteria:

* no informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with clinical diagnosis of HS
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of candidate variants in hair follicles epithelial cell biology by generating Knock-Out (KO) keratinocyte cell lines (HaCaT) | Through study completion, an average of 36 months

SECONDARY OUTCOMES:
Evaluation of the impact of photobiomodulation (PBM) therapy in hair follicles epithelial cells derived from patients and in HaCaT KO cells, | Through study completion, an average of 36 months

CONTACTS AND LOCATIONS:
Locations (15):
- Medical University Innsbruck, Innsbruck, Austria
- Université Libre de Bruxelles, Brussels, Belgium
- France (2):
  - Université Paris Est-Créteil / INSERM U955- Mondor Institute For Biomedical Research (IMRB), Créteil
  - Centre National de la Recherche Scientifique, Strasbourg
- Germany (2):
  - Dessau Medical Cente, Brandenburg
  - Uniklinik Köln, Cologne
- Italy (8):
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinic, Milan
  - Azienda ospedaliero-universitaria pisana, Pisa
  - Istituto Dermopatico dell'Immacolata, IRCCS, Roma
  - Passion people, Roma
  - Policlinico Universitario Fondazione A. Gemelli IRCCS, Roma
  - Ospedale Maggiore di Trieste, Trieste
  - Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste
  - Ospedale San Bortolo, Vicenza
- Jozef Stefan Institute, Ljubljana, Slovenia